CLINICAL TRIAL: NCT00692783
Title: Incidence of Oral Candidiasis, Prevalence of Candida Dubliniensis in HIV Patients and In-vitro Azole Susceptibility. (I.C.O.N.I.C.)
Brief Title: Incidence of Oral Candidiasis, Prevalence of C. Dubliniensis in HIV Patients and In-vitro Azole Susceptibility
Acronym: ICONIC
Status: Terminated | Type: Observational
Why Stopped: Dr. Vindas completed his fellowship + low enrollment
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFJ2008-19
Record Dates: First submitted 2008-05-28; First posted 2008-06-06 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Candidiasis; HIV Infections
Keywords: candida; dubliniensis; candidiasis; HIV; AIDS; azole resistance.
MeSH Terms: conditions — Candidiasis; HIV Infections; Torulopsis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
C. dubliniensis has been identified as pathogen in Oropharyngeal Candidiasis(OPC)particularly among HIV patients. Azole therapy is a cornerstone in OPC, but resistance within C. dubliniensis isolates to diflucan is common.This is a prospective collection of biological specimens from oropharyngeal cavity with the purpose of determining the prevalence of C. dubliniensis in HIV/AIDS patients at the Duval County Department of Health Comprehensive care Center. It is hereto proposed an estimation of azole-resistance in these isolates.

DETAILED DESCRIPTION:
This is a study to try to establish the prevalence of C. dubliniensis as a causative organism of OPC in HIV and/or AIDS patients. We will aim to establish the resistance pattern for azoles but also for Flucytosine and amphotericin of these isolates.

This study will serve as a support to previously published articles that have suggested intrinsic azole-resistance within this particular species of candida and we will try to postulate its possible correlation with clinical failure.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 18 years old or older with a documented diagnosis of HIV infection with or without AIDS-defining illnesses at the time of assessment, who is presenting with clinical symptoms and physical findings compatible with oropharyngeal candidiasis (as defined by the IDSA Guidelines for the Treatment and Management of HIV and HIV- related complications.

Exclusion Criteria:

* Any prior diagnosis or established treatment for oropharyngeal, mucocutaneous or esophageal candidiasis documented in the patient's chart or any proven diagnosis based on reviews of physically available medical records and or history provided by patients that can be subject to later confirmation pertaining to the use of parenteral antifungals within 6 months prior to enrollment (azoles, echinocandins, amphotericin B, Flucytosine, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV with or without AIDS defining illnesses at the Boulevard Comprehensive Care Center
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incidence of oropharyngeal candidiasis in our HIV population; estimation of the prevalence of candida dubliniensis and pattern of azole resistance to direct future treatment | April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jose Vindas, MD, Principal Investigator — University of Florida
Locations (1):
- Duval County Department of Health. Boulevard Comprehensive Care Center, Jacksonville, Florida, United States

REFERENCES:
- [Result] Sullivan D, Coleman D. Candida dubliniensis: characteristics and identification. J Clin Microbiol. 1998 Feb;36(2):329-34. doi: 10.1128/JCM.36.2.329-334.1998. No abstract available. PMID 9466736
- [Result] Milan EP, de Laet Sant' Ana P, de Azevedo Melo AS, Sullivan DJ, Coleman DC, Lewi D, Colombo AL. Multicenter prospective surveillance of oral Candida dubliniensis among adult Brazilian human immunodeficiency virus-positive and AIDS patients. Diagn Microbiol Infect Dis. 2001 Sep-Oct;41(1-2):29-35. doi: 10.1016/s0732-8893(01)00290-5. PMID 11687311
- [Result] Sullivan DJ, Westerneng TJ, Haynes KA, Bennett DE, Coleman DC. Candida dubliniensis sp. nov.: phenotypic and molecular characterization of a novel species associated with oral candidosis in HIV-infected individuals. Microbiology (Reading). 1995 Jul;141 ( Pt 7):1507-21. doi: 10.1099/13500872-141-7-1507. PMID 7551019
- [Result] Sullivan DJ, Moran G, Donnelly S, Gee S, Pinjon E, McCartan B, Shanley DB, Coleman DC. Candida dubliniensis: An update. Rev Iberoam Micol. 1999 Jun;16(2):72-6. No abstract available. PMID 18473572
- [Result] Tintelnot K, Haase G, Seibold M, Bergmann F, Staemmler M, Franz T, Naumann D. Evaluation of phenotypic markers for selection and identification of Candida dubliniensis. J Clin Microbiol. 2000 Apr;38(4):1599-608. doi: 10.1128/JCM.38.4.1599-1608.2000. PMID 10747150
- [Result] Schorling SR, Kortinga HC, Froschb M, Muhlschlegel FA. The role of Candida dubliniensis in oral candidiasis in human immunodeficiency virus-infected individuals. Crit Rev Microbiol. 2000;26(1):59-68. doi: 10.1080/10408410091154183. PMID 10782340